CLINICAL TRIAL: NCT02181153
Title: GENETIC, SEROLOGICAL, FECAL AND CLINICAL MARKERS IN SIBLINGS OF CHILDREN WITH INFLAMMATORY BOWEL DISEASE
Brief Title: Genetic, Serological Fecal and Clinical Markers in Siblings of Children With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Marina Aloi, Assistant Professor, University of Roma La Sapienza
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 01072014
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Inflammatory Bowel Disease
Keywords: inflammatory bowel disease; siblings
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- siblings of patients with IBD (Other): Blood and fecal samples from 100 siblings of children affected with IBD will be collected at the day of enrolment. Clinical risk factors for IBD will be also recorded in a case report form.
  Interventions: Other: sample blood and fecal collection
- patients without family history of IBD (Other): Blood and fecal samples of 100 healthy children without a family history of IBD will be collected at the day of enrolment. Clinical risk factors for IBD will be also recorded in a case report form
  Interventions: Other: sample blood and fecal collection

INTERVENTIONS:
Other: sample blood and fecal collection — Blood and fecal samples will be collected at the day of enrolment

SUMMARY:
Although the precise etiology of inflammatory bowel disease (IBD) is still unknown, over the last decade active research allowed to gain more precise insights in the pathophysiology of IBD indicating that the chronic inflammation of the intestinal mucosa is directed against the microbiota of the gut in particularly susceptible individuals. Genetic studies and more recently genome-wide association studies (GWAS) have allowed to identify over 70 susceptibility genes which confer an increased risk of developing IBD. In the last years the attention of researchers has shifted to the identification of the early immunological changes that occur already at a preclinical stage of the disease, trying also at identifying the disease before it shows itself. Recently, the ability of a combination of serological markers in predicting the development of IBD has been demonstrated in adults. However, there are no studies evaluating a cohort of children at high risk for the disease, in whom the first immunological changes underlying the development of IBD could be studied, including a combination of genetic, serological, fecal and clinical markers.

The purpose of this study is to evaluate in a population genetically well-characterized, as siblings and twins of patients affected with IBD, early genetic, serologic, fecal and clinical markers of disease, which may be present even years before developing the disease. The identification of these markers in predisposed individuals could help to implement strategies for prevention or early treatment to modify the natural history of IBD.

DETAILED DESCRIPTION:
This is a multicenter, prospective, study evaluating the role of serological, genetic, fecal and clinical markers in predicting the development of IBD in a high risk population. The study will be divided in two phases. In the first phase the prevalence of genetic, serologic, fecal, clinical risk factors in 100 siblings of children affected with IBD compared to 100 healthy children with no family history for IBD will be evaluated. The estimated duration of the first phase of the study is 12 months. In a second phase, a long-term follow-up (5 years) will be performed in order to evaluate the accidental cases of IBD in this population.

ELIGIBILITY:
Inclusion Criteria:

* siblings of children affected with IBD
* children without a family history of IBD

Exclusion Criteria:

* age > 18 years
* age < 6 years
* concomitant autoimmune disorders

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the prevalence of known susceptibility genes for IBD in siblings and twins of patients affected with IBD, compared to controls | one year
To evaluate the prevalence of serological markers of autoimmunity known as risk factors for IBD in siblings and twins of patients affected with IBD, compared to controls | one year

SECONDARY OUTCOMES:
To evaluate the presence and values of fecal markers of colonic inflammation in siblings and twins of patients affected with IBD, compared to controls | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Sapienza University of Rome, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Yes